CLINICAL TRIAL: NCT06386783
Title: Fentanyl Versus Dexmedetomidine as an Adjuvant to Bupivacaine in Spinal Anaesthesia for Appendectomy Patients; Peritoneal Symptomatic Effects: A Randomized Clinical Trial
Brief Title: Fentanyl Versus Dexmedetomidine as an Adjuvant to Bupivacaine in Spinal Anesthesia ; Peritoneal Symptomatic Effects
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Soudy Salah Hammad, Lecturer of anesthesia and surgical intensive care, Aswan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Asw.U./823 /7/23
Record Dates: First submitted 2024-04-04; First posted 2024-04-26 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Dexmedetomidine; Fentanyl
Keywords: Peritoneal symptoms; Spinal ansthesia; Appendectomy
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This randomized double blinded study will be conducted at Aswan university hospitals at patients scheduled for emergency appendectomy
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: concealed based on study drugs assigned to each group & to conduct this double -blinded clinical trials, our study drugs will be prepared by the senior anesthesiologist who won't be involved in further observations of the patients and neither patients nor outcome assessor will be aware of which drugs they will receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group D (N.74) (Active Comparator): 5µg Dexmedetomidine {precedexTM 200U/2ml Hospira, Inc,lake forest,iL,USA} (5 µg added by taking 50 µg in a insulin syringe) + 4ml 0.5% heavy bupivacaine HCl.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Group F (N.74) - (Active Comparator): 25 µg Fentanyl {fentanyl Hameln 50 u/ml Gmbh-germany} + 4ml 0.5% heavy bupivacaine HCl.
  Interventions: Drug: Fentanyl HCl

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — Compare between the efficacy of dexmedetomidine and fentanyl as adjuvants on decreasing the intraoperative peritoneal symptoms such as abdominal discomfort or visceral pain, nausea and vomiting, vagal symptoms like bradycardia and hypotension during appendectomy.
  Arms: Group D (N.74)
Drug: Fentanyl HCl — Compare between the efficacy of dexmedetomidine and fentanyl as adjuvants on decreasing the intraoperative peritoneal symptoms such as abdominal discomfort or visceral pain, nausea and vomiting, vagal symptoms like bradycardia and hypotension during appendectomy.
  Arms: Group F (N.74) -

SUMMARY:
To compare whether 5 μg dexmedetomidine with 25 μg fentanyl added to 0.5% hyperbaric bupivacaine as adjuvants in spinal anaesthesia in patients undergoing appendectomy could reduce intraoperative peritoneal related symptoms.

DETAILED DESCRIPTION:
Acute appendicitis is among the most common causes of lower abdominal pain leading patients to attend the emergency department and the most common diagnosis made in young patients admitted to the hospital with an acute abdomen .

In intracavitary abdominal surgery (e.g. Appendectomy),general anesthesia is conventionally chosen as it provides a higher safety profile with respect to the risk of aspiration, abdominal discomfort, and better exposure secondary to muscle relaxation however, at present it is considered safe to do spinal anesthesia in various abdominal procedures, even where significant muscle relaxation is required in certain complex cases such as peritonitis many patients with complicated conditions were operated under spinal anesthesia, which did not significantly interfere with surgical technique or exposure. Additional advantages of spinal anesthesia include faster recovery, better oral tolerance, and shorter hospital stay compared to general anesthesia.

The Covid-19 pandemic currently affects almost every aspect of healthcare. The risk to the operating room team from the contaminated aerosols produced by intubation and positive pressure ventilation may be reduced by performing suitable open operations with neuraxial anaesthesia instead of General anesthesia .

Neuroaxial anesthesia is commonly preferred for surgeries of lower abdomen, perineal and lower limb. It is easy to administer and very economical but needs skills. Intrathecal local anesthetics are limited by short duration of action and needs early use of rescue analgesia postoperatively. Adjuvants are added to improve quality and duration, provide better postoperative analgesia and patient comfort.

A common problem during abdominal surgeries under spinal anesthesia is peritoneal related symptoms as visceral pain, nausea, vomiting, vagal symptoms like bradycardia and hypotension.

Many adjuvants like fentanyl, morphine, ketamine, neostigmine, and clonidine are being used to prolong the analgesic effects of local anaesthetic for many years. These drugs including opioids are usually results in several side effects include itching, decrease respiratory rate, difficulty in urination, postoperative gastrointestinal disturbance which can be overcome by preferring them as adjuvant with other analgesics.

Intraoperative peritoneal related symptoms as visceral pain, nausea, vomiting, vagal symptoms like bradycardia and hypotension are a common problem and there are some intrathecal adjuvants can solve these symptoms.

Fentanyl is µ receptor agonist 80 times more potent than morphine as an analgesic added to spinal 0.5% heavy bupivacaine improves quality of spinal analgesia, reduces visceral and somatic pain. However, their addition may have side effects like pruritus, respiratory depression, urinary retention, postoperative nausea and vomiting which limits their use.

Dexmedetomidine is highly selective α2-agonist, S-enantiomer of veterinary sedative medetomidine. Food and Drug Administration has approved its use for short-term ICU sedation, it is reported to provide sedation that parallels natural sleep, anxiolysis, analgesia, sympatholytic, and anaesthetic-sparing effect with minimal respiratory depression. α2- agonists produce clinical effects.

It was reported in a previous study that intraoperative dexmedetomidine can reduce the incidence of postoperative nausea and vomiting (PONV)in patients undergoing thoracic surgery and a dose-response relationship between intraoperative dexmedetomidine and PONV was Observed; and the optimal dose range for antiemetic effects of PONV is 50-100 μg. Previous small Some meta-analyses demonstrated that intraoperative dexmedetomidine significantly lowered post-operative pain scores and opioid consumption, which could lead to a reduced opioid-related adverse events, including PONV.

Dexmedetomidine prevents and reduces peritoneal related symptoms Intraoperative, and it can significantly lower the demand for opioids and inhalation anesthesia during and after operation, which could help to reduce opioid-related adverse events, including PONV.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status class I and II.
2. Age between 18 - 60 years of either sex.

Exclusion Criteria:

1. ASA grade III and IV.
2. Infection at the site of injection.
3. Coagulopathy or anticoagulation.
4. Congenital anomalies of lower spine.
5. Active disease of CNS.
6. History of allergy to local anesthetics or the adjuvants.
7. Complicated appendicitis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
intraoperative peritoneal symptoms during appendectomy. | Intraoperative period in minutes
  Compare between the efficacy of dexmedetomidine and fentanyl as adjuvants on decreasing the intraoperative peritoneal symptoms such as abdominal discomfort or visceral pain, nausea and vomiting, vagal symptoms like bradycardia and hypotension during appendectomy.

SECONDARY OUTCOMES:
Assessment of motor block with Modified Bromage scale | 1,6,12,18 and 24 hours
  Assessment of motor block with Modified Bromage scale;
  Bromage Scale:
  1. Bromage 0 - patient can move the hip, knee, and ankle.
  2. Bromage 1 - patient is unable to move the hip but can move the knee and ankle.
  3. Bromage 2 - patient is unable to move the hip and knee but able to move the ankle.
     * Onset of Bromage 3 (min), Regression to bromage 0 (min).
  Bromage Scale:
  1. Bromage 0 - patient can move the hip, knee, and ankle.
  2. Bromage 1 - patient is unable to move the hip but can move the knee and ankle.
  3. Bromage 2 - patient is unable to move the hip and knee but able to move the ankle.
Degree of post-operative analgesia | 1,6,12,18 and 24 hours
  VI. The postoperative pain score will be assessed using visual analogue scale (VAS; scored from 0-10, where 0=no pain and 10=the worst pain imaginable) during the recovery room(T0) and at 1,6,12,18 and 24 hours (T1, T6, T12,T18 and T24) in the postoperative period
Assessment of sensory block by using pin prick method | Time in minutes
  Assessment of sensory block by using pin prick method; Time from injection to T10(min) and Time from injection to highest Sensory cephalad spread, Resolution to T10 (min)

CONTACTS AND LOCATIONS:
Overall Officials: Ayman M Eldemrdash, MD, Principal Investigator — Aswan University; Ahmed A Mahmoud, MD, Principal Investigator — Aswan University
Locations (1):
- Aswan University, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minagar M, Alijanpour E, Jabbari A, Rabiee SM, Banihashem N, Amri P, Mir M, Hedayati Goodarzi MT, Esmaili M. The efficacy of addition of dexmedetomidine to intrathecal bupivacaine in lower abdominal surgery under spinal anesthesia. Caspian J Intern Med. 2019 Spring;10(2):142-149. doi: 10.22088/cjim.10.2.142. PMID 31363392
- [Background] Gupta R, Verma R, Bogra J, Kohli M, Raman R, Kushwaha JK. A Comparative study of intrathecal dexmedetomidine and fentanyl as adjuvants to Bupivacaine. J Anaesthesiol Clin Pharmacol. 2011 Jul;27(3):339-43. doi: 10.4103/0970-9185.83678. PMID 21897504